CLINICAL TRIAL: NCT06761378
Title: Ideal Time of Stenting Prior to Ureteral Access Sheath for Stone Disease , Two vs Four Weeks Prospective Study
Brief Title: Ideal Time of Stenting Prior to Ureteral Access Sheath for Stone Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hossam Kandeel, Assistant lecturer of urology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5/2024UROL2
Record Dates: First submitted 2024-12-24; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Ureteric Stone
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Intervention Model Description: Patients and methods The study will be conducted at the urology departments at Menoufia University hospitals. Inclusion criteria: - All patients with stone kidney up to 2 cm, failed ESWL , difficult PCNL Exclusion criteria: - Size more than 2 cm Preoperative assessment by ✓ Full History • personal history ( name ,age ,sex ,residence , occupation , special habits ) • complain • past medical • Past surgical history • family history ✓ Investigations including - laboratory investigations(urine analysis ,CBC ,PT ,AST ,ALT ,Urea, S.creatinine, RBS - Imaging ( CT Urography , KUB) Operative : - Stenting either two weeks or four weeks - Feasibility of Usage of axis sheath - Operative Time - Stone residual - Stent postoperative Disposable flexible URS - Durability - Cost effectiveness Post operative : - complications
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 weeks Dj insertion (Active Comparator): Renal stent for 2 weeks prior flexible uretroscopy
  Interventions: Procedure: Renal stent; Device: Flexible uretroscopy
- 4weeks Dj insertion (Active Comparator): Renal stent for 4 weeks prior flexible uretroscopy
  Interventions: Procedure: Renal stent; Device: Flexible uretroscopy

INTERVENTIONS:
Procedure: Renal stent — Renal stent before flexible uretroscopy
Device: Flexible uretroscopy — Renal stent for 2 weeks prior flexible uretroscopy

SUMMARY:
The miniaturization of endourological instruments and improvements in laser lithotripsy have revolutionized the approach to renal stones . - Flexible URS has become popular with urologists, as it is easy to learn, is associated with high stone-free rates, and is acceptable to patients. Firstly described in 1964 by Marshall, the uretroscope was only passively deflectable and did not include working channel. - Although the first successful procedure in humans with a ureteroscope integrating active deflection has been reported by Takayasu, it was not until 1987 that Demetrius Bagley introduced flexible ureteroscopy as we know it today ).] - two types of flexible uretroscopy can be distinguished : fiberoptic and digital flexible URS. The difference between them is the image relay and light transmission. - Now either to use ureteral access sheath (AS) or not , but usage of AS decrease intrarenal pressure and clear vision by drainage of dust , so , for access of AS stent better to be inserted prior to the procedure ) So, there are little publications regarding the optimal timing of the stent In this study we will assess the feasibility of passage AS after two versus four weeks from stent insertion

DETAILED DESCRIPTION:
The miniaturization of endourological instruments and improvements in laser lithotripsy have revolutionized the approach to renal stones . - Flexible URS has become popular with urologists, as it is easy to learn, is associated with high stone-free rates, and is acceptable to patients. Firstly described in 1964 by Marshall, the uretroscope was only passively deflectable and did not include working channel. - Although the first successful procedure in humans with a ureteroscope integrating active deflection has been reported by Takayasu, it was not until 1987 that Demetrius Bagley introduced flexible ureteroscopy as we know it today ).] - two types of flexible uretroscopy can be distinguished. The difference between them is the image relay and light transmission. - Now either to use ureteral access sheath (AS) or not , but usage of AS decrease intrarenal pressure and clear vision by drainage of dust , so , for access of AS stent better to be inserted prior to the procedure ) So, there are little publications regarding the optimal timing of the stent In this study we will assess the feasibility of passage AS after two versus four weeks from stent insertion

ELIGIBILITY:
Inclusion Criteria:

* All patients with stone kidney up to 2 cm
* failed ESWL (extracorporeal shock wave lithotripsy)
* difficult PCNL (percutaneous nephrolithotomy)

Exclusion Criteria:

* Size more than 2 cm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
passage of access sheath after dilation of the ureter by DJ 2 vs 4 weeks | 6 months
  Patients will classified in two groups, one will insert DJ for two weeks and the other insert DJ for four weeks then remove it and trial to insert access sheath for flexible uretroscopy duriing passage of the sheath the ureteric dilitation will be assessed if the sheath pass or not measure so , the ability of the ureteric dilitation to obtain the sheath is it dilated enough after 2 or 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Menofia university, Cairo, State Or Province, Egypt